CLINICAL TRIAL: NCT01115621
Title: BABYDIET-Study - Primary Prevention of Type 1 Diabetes in Relatives at Increased Genetic Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut fur Diabetesforschung, Munich, Germany (Other)
Responsible Party: Prof. Dr. Anette-G. Ziegler, Institut fuer Diabetesforschung, Ingolstädter Landstr. 1, Neuherberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZI310/14-1
Record Dates: First submitted 2010-04-07; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutenfree diet (Active Comparator): Glutenfree diet during the first year of life
  Interventions: Other: Glutenfree diet during the first year of life
- Control - normal diet (No Intervention)

INTERVENTIONS:
Other: Glutenfree diet during the first year of life — Glutenfree diet during the first year of life
  Arms: Glutenfree diet

SUMMARY:
The major goals of this project are to determine whether primary intervention through delayed introduction of dietary gluten is feasible and could reduce the incidence of islet autoimmunity in high-risk first degree relatives of patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Newborn offspring or siblings of patients with type 1 diabetes with a HLA genotype conferring a high diabetes risk

Exclusion Criteria:

* If infants have an illness or birth defect that precludes long-term follow-up or involves use of treatment that may alter the natural history of diabetes

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2001-02; Primary Completion 2009-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effect of dietary intervention on the development of islet autoantibodies | 3 years
  Primary outcome is to compare the prevalence of iselt autoantibodies between children participating in the dietary intervention and the control group.

SECONDARY OUTCOMES:
Effect of dietary intervention on the development of Type 1 diabetes. | 10 years
  Secondary outcome is to compare the prevalence of type 1 diabetes between children participating in the dietary intervention and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Anette G Ziegler, MD, Principal Investigator — Institut für Diabetesforschung, München, Germany
Locations (1):
- Institut für Diabetesforschung, München, Germany

REFERENCES:
- [Background] Winkler C, Hummel S, Pfluger M, Ziegler AG, Geppert J, Demmelmair H, Koletzko B. The effect of maternal T1DM on the fatty acid composition of erythrocyte phosphatidylcholine and phosphatidylethanolamine in infants during early life. Eur J Nutr. 2008 Apr;47(3):145-52. doi: 10.1007/s00394-008-0708-9. Epub 2008 Apr 28. PMID 18443841
- [Background] Pfluger M, Winkler C, Hummel S, Ziegler AG. Early infant diet in children at high risk for type 1 diabetes. Horm Metab Res. 2010 Feb;42(2):143-8. doi: 10.1055/s-0029-1241830. Epub 2009 Nov 9. PMID 19902403
- [Result] Schmid S, Buuck D, Knopff A, Bonifacio E, Ziegler AG. BABYDIET, a feasibility study to prevent the appearance of islet autoantibodies in relatives of patients with Type 1 diabetes by delaying exposure to gluten. Diabetologia. 2004 Jun;47(6):1130-1. doi: 10.1007/s00125-004-1420-9. Epub 2004 May 28. No abstract available. PMID 15168019
- [Derived] Laimighofer M, Lickert R, Fuerst R, Theis FJ, Winkler C, Bonifacio E, Ziegler AG, Krumsiek J. Common patterns of gene regulation associated with Cesarean section and the development of islet autoimmunity - indications of immune cell activation. Sci Rep. 2019 Apr 18;9(1):6250. doi: 10.1038/s41598-019-42750-5. PMID 31000755
- [Derived] Hummel S, Pfluger M, Hummel M, Bonifacio E, Ziegler AG. Primary dietary intervention study to reduce the risk of islet autoimmunity in children at increased risk for type 1 diabetes: the BABYDIET study. Diabetes Care. 2011 Jun;34(6):1301-5. doi: 10.2337/dc10-2456. Epub 2011 Apr 22. PMID 21515839
- [Derived] Adler K, Mueller DB, Achenbach P, Krause S, Heninger AK, Ziegler AG, Bonifacio E. Insulin autoantibodies with high affinity to the bovine milk protein alpha casein. Clin Exp Immunol. 2011 Apr;164(1):42-9. doi: 10.1111/j.1365-2249.2011.04324.x. Epub 2011 Mar 1. PMID 21361910